CLINICAL TRIAL: NCT07328763
Title: The Effect of Pranayama Breathıng Exercıses on Paın, Anxıety,aAnd Sleep Qualıty in Indıvıduals wıth Fıbromyalgıa
Acronym: Pranayama
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ondokuz Mayıs University (Other)
Responsible Party: Principal Investigator, Aybike Kose, Registered Nurse (RN), Ondokuz Mayıs University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2025/224
Record Dates: First submitted 2025-12-19; First posted 2026-01-09 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2025-12

CONDITIONS: Patients Diagnosed With Fibromyalgia Syndrome
Keywords: Fibromyalgia, Nursing, Pranayama, Quality of Life, Anxiety, Sleep Quality
MeSH Terms: conditions — Fibromyalgia; Anxiety Disorders; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Intervention Model Description: The study used block randomization. Block randomization was performed by an independent researcher. In the randomization, two different groups were coded with different letters (A, B) and blocks were formed. Then, random numbers were assigned to the blocks using a computer. The letters assigned in the randomization were written in sealed envelopes and kept. After identifying patients who met the inclusion criteria, informed consent was obtained, pre-tests were administered, and then the independent researcher was contacted to determine which group the patient belonged to. Patients diagnosed with fibromyalgia who present to the polyclinic will be referred to the researcher. Before starting the study, informed consent will be obtained from the participating patients. Patients in the control group will be given an appointment schedule including their scheduled dates. Patients in the experimental group will have an exercise plan developed and will be given an appointment schedule including
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Patients in the control group will be given an appointment schedule containing their scheduled interview dates.
- Pranayama (Experimental): Pranayama breathing exercises will be taught online for 20 minutes, twice a week for 6 weeks.
  Interventions: Other: Pranayama breathing exercises

INTERVENTIONS:
Other: Pranayama breathing exercises — Step 1: Normal breathing, focusing on the breath Step 2: Sun Breath (Surya Prana) Step 3: Alternate Nose Breathing (Nadi Shodhana) Step 4: Ocean Breath (Ujiayi) Step 5: Normal breathing, focusing on the breath
  Arms: Pranayama

SUMMARY:
Individuals diagnosed with fibromyalgia syndrome have a low quality of life due to factors such as pain, sleep problems, high anxiety, depression and low self-esteem, difficulty performing daily living activities, and inhibited socialization (García-Martínez et al., 2012; Sieczkowska et al., 2020). Nurses apply care with a holistic approach philosophy that includes supportive, preventive, therapeutic, and rehabilitative aspects to promote and maintain health. Pranayama is an effective, non-invasive, cost-effective, and easily applicable approach that can be implemented within the framework of holistic care (İlter & Ovayolu, 2021). It is the nurse's responsibility to provide care and create a comfortable environment for patients, improving their quality of life (Aktaş & İlgin, 2023). In this regard, during the application and teaching of breathing exercises, nurses should carefully assess patients' belief in these exercises. They should plan with the patient the appropriate time, duration, and environment for breathing exercises and be able to evaluate the results (ÖZ, 2020). Studies evaluating the results of applying pranayama to individuals with fibromyalgia are limited in the literature. Therefore, it is thought that pranayama could greatly facilitate and provide concrete data on improving the quality of life for individuals with fibromyalgia by reducing pain, sleep problems, anxiety, and improving functionality.

DETAILED DESCRIPTION:
Fibromyalgia syndrome (FMS) is a rheumatological syndrome characterized by symptoms such as increased pain sensitivity, sleep disturbances, fatigue, musculoskeletal pain, stiffness, tenderness, cognitive dysfunction, and mood disorders due to dysregulation of neurophysiological functions (Singh & Rao, 2023; Verma et al., 2020). The incidence of FMS in the general population is reported to be 2-8%, predominantly affecting women (between 61% and 90%), with a male/female ratio of 2.3 (Galvez-Sánchez et al., 2019; Jones et al., 2015; Schmidt-Wilcke & Diers, 2017). Although there are insufficient prevalence studies in Turkey, a study conducted in the Trabzon region found the prevalence of FMS to be 3.6% in women aged 20-64 and 0.9% in women aged 20-29 (Topbas et al., 2005).

The American College of Rheumatology (ACR) first defined the FM Diagnostic Criteria in 1990, and these criteria were revised in 2010, 2011, and 2016 (Plesner & Vaegter, 2018). While there is no definitive treatment method, pharmacological and non-pharmacological treatment methods are applied. Non-pharmacological treatments include acupuncture, biofeedback, capsaicin, chiropractic, cognitive behavioral therapy, exercise, hydrotherapy, spa therapy, massage, meditative movement (Qigong, yoga, and Tai Chi), mindfulness/mind-body therapy, multicomponent therapy, and S-adenyl methionine. In addition, methods such as physical therapy, stretching, strengthening, aerobic exercise, and endurance training are also used (Chitra et al., 2017; Prabhakar et al., 2019).

Fibromyalgia is a common disease associated with numerous comorbidities and is often difficult to diagnose, which can have a devastating impact on quality of life, impair patients' abilities, lead to social and psychological problems for patients, and create a significant socioeconomic burden on healthcare systems (Atahan et al., 2023; Kang et al., 2022).

Fibromyalgia presents with chronic pain without any apparent peripheral tissue damage. This pain results from threatening tissue damage that activates peripheral nociceptors without real or definitive evidence (Ruschak et al., 2023). The pain is characterized by morning stiffness and increasing intensity throughout the day, is anatomically widespread, and is accompanied by hyperexcitability with increased response of the central nervous system to various stimuli (pressure, temperature, light, and medication, etc.). It is characterized by hyperalgesia, allodynia, and features reflected in multiple spinal segments (Araya-Quintanilla et al., 2020).

Patients with FM syndrome may experience emotionally impactful situations in the form of high levels of stress, anger, and catastrophic scenario-based pain, and these situations can worsen existing symptoms (Galvez-Sánchez et al., 2019). Studies have reported that a significant proportion of FM patients experience depression, panic disorder, and anxiety disorder (Basar et al., 2023; Siracusa et al., 2021). It is thought that the cognitive and psychological processes experienced by patients are related to pain (Cetingok et al., 2022). One study reported that FS patients were more likely to experience depression (20%-80%) and anxiety (13%-63.8%) (Henao-Pérez et al., 2022). A meta-analysis study suggested that the lifetime prevalence of depression in fibromyalgia is approximately 65% (Galvez-Sánchez et al., 2020).

Sleep problems are one of the factors triggered by pain and impairing quality of life in individuals diagnosed with fibromyalgia (FS) (Choy, 2015; Keskindag & Karaaziz, 2017). One study reported that poor sleep quality was perceived as a serious symptom in patients diagnosed with FS, negatively impacting multiple health-related symptoms such as pain, fatigue, cognitive complaints, poor functionality, and low work performance (Climent-Sanz et al., 2020). Another study found that compared to healthy individuals, individuals diagnosed with FS had significantly higher numbers of awakenings, awakening index, and sleep apnea syndrome, and poor sleep quality (Çetin et al., 2020). Pranayama involves the control of breath, a dynamic bridge between body and mind. In Sanskrit, "Pranayama" is a combination of the words "Prana" and "ayama." Prana means breath, vitality, life, and energy, while ayama means restriction, control, or regulation. Pranayama can be described as 'the science of breath, breath control, willful breathing' (İlter & Ovayolu, 2021). The breathing cycle in pranayama consists of three stages: Puraka (inspiration), Rechaka (expiration), and Kumbhaka (inhalation and holding the breath after inhalation) (İyengar, 2022).

Recent studies have shown that pranayama, by providing body and mind control, contributes to the improvement of many symptoms of fibromyalgia (Singh & Rao, 2023). Pranayama has been reported to significantly improve the management of many symptoms of fibromyalgia, including pain intensity, stiffness, anxiety, stress, low muscle strength, fatigue, sleep problems, as well as flexibility and cognition, and to improve quality of life (Chitra et al., 2017; Firestone et al., 2014; Hennard, 2011; Lazaridou et al., 2019; Verma et al., 2020). This research was designed as a pre-test-post-test, randomized controlled, experimental study to determine the effects of pranayama breathing exercises on pain, anxiety, sleep quality, and overall health status in individuals with fibromyalgia.

Research Objectives and Hypotheses This research was planned to determine the effects of pranayama breathing exercises applied to individuals with fibromyalgia on pain, anxiety, sleep quality, and health status.

H1: Pranayama breathing exercises applied to individuals with fibromyalgia have an effect on pain. H2: Pranayama breathing exercises applied to individuals with fibromyalgia have an effect on anxiety.

ELIGIBILITY:
Inclusion Criteria:

* Individuals aged 18 and over,
* having experienced pain for at least three months,
* diagnosed with fibromyalgia by a physician according to the ACR 2016
* romyalgia diagnostic criteria,
* having a PUKI score of five or higher,
* having a VAS pain score of one or higher,
* having no communication problems,
* and not being pregnant.

Exclusion Criteria:

* Individuals with a history of respiratory diseases such as malignancy or tuberculosis,
* those with a psychiatric diagnosis,
* those with nasal obstruction due to septal deviation,
* and those who have previously participated in a similar breathing exercise program will be excluded from the study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2025-06-01 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-01-30 (Estimated)

PRIMARY OUTCOMES:
Visual Analog Scale (VAS) | 6 Weeks
  To indicate the severity of your pain, place an (I) mark on one of the lines below. 0 points: no pain, 1-2 points: very mild pain, 3-4 points: mild pain, 5-6 points: moderate pain, 7-8 points: severe pain, 9-10 points: very severe pain.
Pittsburgh Sleep Quality Index (PSQI) | 6 Weeks
  questions only relate to habits from the past month.
Beck Anxiety Scale (BAS) | 6 Weeks
  Some symptoms that people experience when they are anxious or worried.
Fibromyalgia Impact Questionnaire (FIQ) | 6 Weeks
  Severity of fibromyalgia symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Aybike KÖSE, Principal Investigator — Samsun Provincial Health Directorate
Locations (1):
- Samsun Physical Medicine and Rehabilitation Hospital, Samsun, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
The sample group participating in the study gave their consent for the information not to be shared.